CLINICAL TRIAL: NCT06495736
Title: Application of Rapid On-site Evaluation in Lymph Node Biopsy of Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yunnan Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024.76
Record Dates: First submitted 2024-06-25; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Histology Paraffin dyeing (No Intervention)
- ROSE technique (Experimental)
  Interventions: Diagnostic Test: Experimental: ROSE technique stain
- Cytological HE staining (No Intervention)
- Cytological Pap staining (No Intervention)

INTERVENTIONS:
Diagnostic Test: Experimental: ROSE technique stain — The ROSE technical group uses Diff-Quick stain for diagnosis
  Arms: ROSE technique

SUMMARY:
The goal of this clinical trial is to evaluate the value of rapid on-site evaluation（ROSE） in lymph node biopsy of breast cancer. The main question it aims to answer is:The ROSE technique was applied to breast cancer lymph node biopsy to improve the diagnostic efficiency and accuracy.

Participants underwent routine lymph node biopsy, and the test personnel conducted routine disease examination and rose technique evaluation on the removed ly

ELIGIBILITY:
Inclusion Criteria:

* Patients had pathologically confirmed primary breast cancer
* Surgical treatment was available

Exclusion Criteria:

* Previous history of surgery on the affected axilla, internal breast or chest
* Pregnant or breastfeeding patients
* Previous radiotherapy or chemotherapy
* Complicated history of other tumors

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
The number of positive and negative lymph nodes diagnosed by ROSE technique | up to 2 years

SECONDARY OUTCOMES:
The time taken to diagnose using the ROSE technique | up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Yunnan Cancer Hospital, Kunming, Yunnan, China